CLINICAL TRIAL: NCT07112326
Title: Evaluating Community Gardens as Environmental Health Interventions in Mississauga
Brief Title: Community Gardens and Environmental Health in Mississauga
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Vasanti Malik, Associate Professor, University of Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 48687
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes
Keywords: community gardening; type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: One-group pretest-posttest design involving:
  1. Participation in Ecosource's 26-week community garden program.
  2. Evaluating the program's impact on type 2 diabetes risk factors, including diet quality and physical activity, and its alignment with Mississauga's Healthy City Strategy by improving access to healthy foods and green spaces, through surveys at at baseline, 12 weeks, and 26 weeks, assessing diet quality
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Participation in Ecosource's 26-week community gardening and cooking classes with nutrition and type 2 diabetes education
  Interventions: Behavioral: Community Gardening Program

INTERVENTIONS:
Behavioral: Community Gardening Program — Participants will take part in a 26-week community gardening program with Ecosource, which involves cooking classes, as well as nutrition and type 2 diabetes education. These weekly sessions will be led by Ecosource and take place in community gardens across different sites in Mississauga and at Ecosource's teaching kitchens. Diabetes education sessions will take place once per month (6 times/program) and will be led by subject matter experts including dietitians/diabetes educators. The delivery format for these sessions may be virtual or in-person depending on the topic covered and participant availability. Participants will be invited to a WhatsApp Community Chat to stay motivated and engaged with the study over the 26-week period.

SUMMARY:
The goal of this clinical trial is to evaluate a revised version of Ecosource's 26-week community garden program. This project aims to assess how community gardening can reduce type 2 diabetes risk and improve health outcomes among people aged 18 and older, who have type 2 diabetes, type 2 diabetes risk factors, or interest in type 2 diabetes prevention. The project's objectives are to:

1. Co-design and deliver a revised 26-week program integrating type 2 diabetes education into Ecosource's community garden program.
2. Evaluate the program's impact on type 2 diabetes risk factors, including diet quality and physical activity, and its alignment with Mississauga's Healthy City Strategy by improving access to healthy foods and green spaces.
3. Share findings to inform future community gardening initiatives aimed at reducing type 2 diabetes risk and promoting health.

Participants will:

* Participate in a co-design focus group
* Complete 3 questionnaires about diet quality and T2D risk factors at baseline, 12 weeks, and 26 weeks.
* Participate in a photovoice project and focus group
* Participate in a post-implementation focus group

DETAILED DESCRIPTION:
Ecosource's community garden program is highlighted in Mississauga's Healthy City Strategy as a key initiative to enhance access to affordable, healthy food at the neighbourhood level. With food insecurity increasing in Mississauga-evidenced by a 58% increase in visitors to the city's largest food bank from June 2023 to May 2024 and the subsequent declaration of a food insecurity emergency by City Council-urgent interventions are needed. Additionally, demand for community gardening has reached unprecedented levels, with over 2,000 people on the waitlist, a trend likely exacerbated by rising housing and food costs. Food insecurity is also a known risk factor for type 2 diabetes making the case for initiatives that address food access as a health promotion strategy. A healthful diet and lifestyle are the cornerstones of chronic disease prevention. Community gardening programs have emerged as a strategy to improve diet quality especially when paired with nutrition education. In addition, Ecosource's program has a proven history of engaging residents, including in priority neighbourhoods where type 2 diabetes prevalence exceeds the provincial average. The majority of Ecosource's garden sites are in public parks within these communities, including Malton and areas along the western Hurontario corridor. Gardens in these areas have some of the longest waitlists across our network, indicating a high interest in gardening in these neighbourhoods. Since 2006, Ecosource has built partnerships to reduce barriers to gardening access, engaging over 17 community partners annually. Survey data from program participants also indicates the program's readiness for further development and evaluation, with findings suggesting gardening offers co-benefits for food access, physical activity, community belonging, and mental health.

Therefore, this project aims to strengthen and evaluate the program's impact on promoting health in priority neighbourhoods, with a focus on type 2 diabetes prevention, while addressing the food insecurity crisis in Mississauga. The Evaluating Community Gardens as Environmental Health Interventions in Mississauga project aims to assess how community gardening can reduce type 2 diabetes risk and improve health outcomes in Mississauga's priority communities. Building on Ecosource's successful community garden program, this project explores community gardening as a strategy for improving diet quality and food access, both linked to type 2 diabetes prevention. The project is timely, given concerns over rising food insecurity following Mississauga's emergency declaration and the inclusion of community gardens in municipal health, food security, and climate resiliency plans.

Goals and Research Aims:

The research team will design, deliver and evaluate a revised version of Ecosource's community garden program, aiming to strengthen its effectiveness in preventing type 2 diabetes and promoting health. The program will engage 20-30 residents from priority areas, such as Malton and western Hurontario, in weekly sessions at Ecosource's gardens and teaching kitchen. The 26-week program will consist of weekly two-hour sessions.

The project's objectives are to:

1. Co-design and deliver a revised 26-week program integrating type 2 diabetes education into Ecosource's community garden program.
2. Evaluate the program's impact on type 2 diabetes risk factors, including diet quality and physical activity, and its alignment with Mississauga's Healthy City Strategy by improving access to healthy foods and green spaces.
3. Share findings to inform future community gardening initiatives aimed at reducing type 2 diabetes risk and promoting health.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years or older.
* Have an interest in Type 2 Diabetes (T2D) prevention OR have a diagnosis of T2D or have risk factors for T2D.
* Should not have any chronic disease that could affect participation in the study
* Not currently participating in another trial/research study (other than the current one)
* Must be a resident of Mississauga

Exclusion Criteria:

* People under 18 years
* Has a Chronic disease that could affect participation in the study
* Currently participating in another trial/research study (other than the current one)
* Not a resident of Mississauga

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-07-02 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Changes in diet quality | Baseline, 12 weeks and 26 weeks
  Changes in diet quality will be assessed according to the Canadian Food Intake Screener. The questions in this screener ask participants about foods and beverages they ate or drank in the past 30 days. The Canadian Food Intake Screener is a tool used to assess the alignment of a person's eating habits with the recommendations of Canada's Food Guide. The total score, which can range from 0 to 65, reflects the degree of alignment with healthy eating recommendations.

SECONDARY OUTCOMES:
Changes in physical activity | Baseline, 12 weeks and 26 weeks
  Participants will be asked to complete a questionnaire that includes questions from the International Physical Activity Questionnaire. These questions will collect information about the physical health and activity of the participant, which will help the researchers determine the impact of exercise and physical activity on type 2 diabetes risk factors.
Food literacy | Baseline, 12 weeks and 26 weeks
  The researchers will measure food literacy using the the Canadian Behaviour Attitude and Nutrition Knowledge Survey (C-BANKS). This tool is used to assess Canadians' knowledge, attitudes, and behaviors related to nutrition.
Food Security | Baseline, 12 weeks and 26 weeks
  The researchers will use the Household Food Security Survey Module (HFSSM) to measure food security. This is a standardized set of 18 questions used to measure food insecurity in Canadian households. It's the primary tool used in Canada to assess how limited financial resources impact a household's ability to acquire adequate food. The HFSSM categorizes food insecurity into three levels: marginal, moderate, and severe.
Type 2 diabetes risk | Baseline, 12 weeks and 26 weeks
  The researchers will measure type 2 diabetes risk using the Canadian Diabetes Risk Questionniare (CANRISK). This questionnaire assesses an individual's risk of having prediabetes or type 2 diabetes. The questionnaire gathers information on risk factors like age, family history, ethnicity, and lifestyle, and calculates a score indicating the likelihood of having prediabetes or diabetes.
Alignment with Mississauga's Healthy City Strategy | Baseline, 12 weeks and 26 weeks
  The research team will collect additional metrics such as pounds (lbs) of food grown and visits to gardens in priority areas, to assess alignment with Mississauga's Healthy City Strategy.

CONTACTS AND LOCATIONS:
Overall Officials: Vasanti Malik, MSc, ScD, Principal Investigator — University of Toronto
Locations (4):
- Canada (4):
  - Malton Community Garden, Mississauga, Ontario
  - Iceland Teaching Garden, Mississauga, Ontario
  - Ecosource Community Climate Hub, Mississauga, Ontario
  - Parkway Green Generation Garden, Mississauga, Ontario (ON)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-07-02): https://cdn.clinicaltrials.gov/large-docs/26/NCT07112326/ICF_000.pdf